CLINICAL TRIAL: NCT04486742
Title: Brief Cognitive Behavioral Therapy to Treat Itch Rumination "Itch CBT" in Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Amy Paller, Study Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2019-2560
Record Dates: First submitted 2020-07-14; First posted 2020-07-27 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Atopic Dermatitis
Keywords: Pediatric
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itch CBT Arm (Experimental): Participants randomized to the Itch CBT Arm will participate in 4 weekly telehealth sessions with a therapist to address common areas of anxiety related to atopic dermatitis.
  Interventions: Behavioral: Itch CBT
- Usual Care Arm (No Intervention): Participants randomized to the Usual Care Arm of the study will receive standard of care eczema educational materials that are typically provided by their health care provider after a clinic (or telehealth) visit.

INTERVENTIONS:
Behavioral: Itch CBT — Telemedicine CBT sessions with a therapist to address atopic dermatitis related concerns.
  Arms: Itch CBT Arm

SUMMARY:
The main purpose of this study is to adapt cognitive behavior therapy (CBT) to improve itch in children with eczema.

DETAILED DESCRIPTION:
Eczema is characterized by chronic itch. Many children develop a chronic focus (rumination) on their itch. Rumination is a maladaptive method of responding to distress, in which the individual thinks obsessively about the source of distress. The rumination on chronic itch in eczema can have detrimental effects on one's quality of life, as well as induce significant anxiety about when itch will return, how long it will last, and how it will affect physical and social functioning.

Cognitive behavior therapy (CBT) is a frontline treatment for rumination, as it focuses on teaching strategies so that the individual can examine distressing thoughts objectively and determine their validity, replace negative thinking patterns with more adaptive thought patterns, and increase the individual's awareness to their problematic thought patterns. Additionally, CBT helps the individual to implement behavioral strategies to cope with possibly anxiety-inducing situations, such as scratching while trying to go to sleep.

The investigators hypothesize that an Itch CBT intervention is an effective, non-medication-based, easy to implement strategy to improve itch in children with eczema.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe atopic dermatitis [assessed by Patient Oriented Eczema Measure (POEM)score of >-8 OR NRS itch score of >= 4].
* English speaking.
* Currently receiving treatment at Lurie Children's Hospital for atopic dermatitis.
* Parent or guardian available to participate in protocol.
* Have sufficient technology (e.g., cell phone, computer, tablet, etc.) that can be used to access Zoom conference technology for telemedicine visits.

Exclusion Criteria:

* Inability to comprehend and complete questionnaires.
* History of intellectual disability or psychosis.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Itch Severity Numerical Rating Scale | Baseline to Week 4
  Numerical rating scale to assess itch severity, scale of 0-10, higher score means higher itch severity and worse outcome.

SECONDARY OUTCOMES:
Itch Rumination Questionnaire | Baseline to Week 4
  Questionnaire to assess common fear and anxiety around itch
PROMIS Anxiety and Depression | Baseline to Week 4
  Questionnaire to assess anxiety and depression symptoms in pediatric populations
PROMIS Pediatric Itch - Short Form 1 (2+6) | Baseline to Week 4
  Questionnaire to assess level and severity of itch and common disturbances due to itch (social, emotional, physical)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT04486742/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT04486742/ICF_001.pdf